CLINICAL TRIAL: NCT06506474
Title: Low-value Care, and Variation in Practice for Children Hospitalized With Bronchiolitis - a Multicentric Prospective Observational Study
Brief Title: Low-value Care, and Variation in Practice for Children Hospitalized With Bronchiolitis
Acronym: CareBEST
Status: Recruiting | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Maternal Infant Child and Youth Research Network (Unknown); The Hospital for Sick Children (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Olivier Drouin, M.D., M.Sc M.P.H., Pediatrician and Clinical Assistant Professor, Departments of Paediatrics and Department of Social and Preventive Medicine, St. Justine's Hospital
Other Study IDs: 2024-5815
Record Dates: First submitted 2024-05-30; First posted 2024-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Bronchiolitis
Keywords: infants; hospitalization; bronchiolitis; low-value care; observational study
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (15):
- Children admitted to CHU Sainte-Justine: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to McMaster Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to British Columbia Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to IWK Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to CHU de Quebec University Laval Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Montreal Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Children's Hospital of Eastern Ontario: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Kingston Health Sciences Centre: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to The Hospital for Sick Children: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
- Children admitted to Children's Hospital of Western Ontario: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Alberta Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Stollery Children's Hospital: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children Admitted to Hôpital Maisonneuve-Rosemont: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Cité-de-la-Santé: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis
- Children admitted to Lakeridge Health: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis, admitted to a general pediatric inpatient unit, not previously recruited for the study.
  Interventions: Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis

INTERVENTIONS:
Diagnostic Test: Provision of any of six different low-value health services for treatment of bronchiolitis — This prospective observational will have six separate primary outcomes acting as exposures, (or interventions).The exposures are the the provision of any of the six low-value health services: 1) respiratory virus testing; 2) chest x-ray; 3) continuous pulse oximetry; 4) short-acting beta-agonists; 5) systemic corticosteroids; and 6) antibiotics.
  Groups: Children Admitted to Hôpital Maisonneuve-Rosemont; Children admitted to Alberta Children's Hospital; Children admitted to British Columbia Children's Hospital; Children admitted to CHU Sainte-Justine; Children admitted to CHU de Quebec University Laval Hospital; Children admitted to Children's Hospital of Eastern Ontario; Children admitted to Children's Hospital of Western Ontario; Children admitted to Cité-de-la-Santé; Children admitted to IWK Children's Hospital; Children admitted to Kingston Health Sciences Centre; Children admitted to Lakeridge Health; Children admitted to McMaster Children's Hospital; Children admitted to Montreal Children's Hospital; Children admitted to Stollery Children's Hospital

SUMMARY:
Low-value care is defined as the use of a health service, such as diagnostics and treatments, for which the harms or costs outweigh the benefits. In pediatrics, investigations or treatments can be unpleasant or traumatizing to the child, can prolong the time spent in hospital, and can create a cascade of further futile investigations and treatments. Several of the commonly used diagnostics and treatments in bronchiolitis are considered low-value, making it a great model to study low-value care in pediatrics.

The purpose of CareBEST is to study the use of 6 low-value healthcare services in children aged 1 to 12 months hospitalized with bronchiolitis, their costs, and measure the variability in practice of these services.

The main questions this study aims to answer are:

1. How frequently are 6 low-value care health services used in children hospitalized with bronchiolitis? These 6 low-value care health services are: 1) respiratory virus testing; 2) chest x-rays; 3) continuous pulse oximetry; 4) short-acting beta-agonists; 5) systemic corticosteroids; and 6) antibiotics.

   * Are there factors that predict the use of these services?
   * What are the costs of the use of these services?
2. How much variability is there between different patients, different doctors, and between hospitals in the use of these 6 low-value health services ?
3. Are differences in use of low-value health services associated with patient and family characteristics (like race and ethnicity, socioeconomic status, language), and do these contribute to disparities in care?

Participants will have their infant's medical chart reviewed during their hospitalization. They will also have 2 short questionnaires to complete, once during their child's admission to the hospital, and one 30 days later to ask about whether their child required any additional medical care. They will additionally be asked to complete a questionnaire on their perceptions regarding their child's care while hospitalized, including the use of shared-decision making and their understanding of and involvement in the care decisions made.

This analysis will provide a better understanding of treatment of bronchiolitis in Canada and help in the development of effective interventions to reduce low-value care.

DETAILED DESCRIPTION:
Background: Low-value care is defined as the use of a health service, such as diagnostics and treatments, for which the harms or costs outweigh the benefits. Reducing low-value care is important in improving the health of Canadians and achieving a sustainable, high-quality healthcare system. Bronchiolitis is among the most common and most costly causes of hospitalizations in children. Most healthcare costs associated with bronchiolitis are related to hospitalization, and these costs have been increasing. Supportive care is recommended by national guidelines for the treatment of bronchiolitis, and many commonly used diagnostics and treatments in bronchiolitis are considered low-value, making it a great model to study low-value care in pediatrics. To develop effective interventions to reduce low-value care, and ensure the right resources go to the right patient at the right time, it is crucial to develop a better understanding of inpatient management of bronchiolitis in Canada.

The goal of this prospective multi-site observational study is to analyze the use of 6 low-value healthcare services in children diagnosed with bronchiolitis, their costs, and measure the variability in practice of these services.

Specific objectives: Among infants admitted with bronchiolitis at 15 Canadian hospitals with pediatric admissions, to:

1. Measure the incidence, patterns, and predictors of use of 6 low-value care health services and their costs in children hospitalized for bronchiolitis, namely 1) respiratory virus testing; 2) chest x-rays; 3) continuous pulse oximetry; 4) short-acting beta-agonists; 5) systemic corticosteroids; and 6) antibiotics;
2. Estimate the extent of practice variation in the use of 6 low-value health services between hospitals;
3. Determine whether differences in use of low-value health services are associated with patient and family characteristics (e.g., race and ethnicity, socioeconomic status, language), and whether these contribute to disparities in care.

Design: A multi-centre (n=15), prospective observational cohort study of children hospitalized with bronchiolitis. Data will be obtained from medical charts and entered into a central, web-based REDCap database. A health equity questionnaire will be completed by participants once during their child's admission and then again 30 days later to inquire on additional medical care required post-admission. Secondary outcomes and covariates will also be collected which include but are not limited to duration of ICU stay, use of mechanical ventilation, cardiac arrest, length of hospital stay, disease severity, clinician years of experience, and death.

Analysis of the primary outcome will be descriptive for each low-value health service, overall and stratified by sex. Costs of hospitalization will be assessed from a healthcare institution perspective. Cost of each of low-value health service will be described and compared between one another and across sites to identify key differences which may be targets for process change.

This study will provide important data to understand the use of low-value care in bronchiolitis treatment in Canada, and will inform our approach to addressing low-value care in bronchiolitis and in other common conditions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged >28 days to <12 months
* Children admitted to a pediatric inpatient ward with an admission diagnosis of bronchiolitis

Exclusion Criteria:

- Children previously recruited for the study, either during a previous bronchiolitis admission or for the same incident of bronchiolitis, while admitted to another study site.

Ages: 28 Days to 12 Months | Sex: All
Age Groups: Child
Study Population: Children aged >28 days to <12 months with an admission diagnosis of bronchiolitis.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of eligible patients receiving each of the six low-value health services | 24 months
  The primary outcome of the study is the proportion of patients receiving each of the six low-value health services during their hospitalization for bronchiolitis: 1) respiratory virus testing; 2) chest x-ray; 3) continuous pulse oximetry; 4) short-acting beta-agonists; 5) systemic corticosteroids; and 6) antibiotics.

SECONDARY OUTCOMES:
Transfer to the ICU | 24 months
  Whether the child admitted with bronchiolitis was transferred to the ICU. If so, duration of ICU stay.
Use of CPAP, BiPAP, or mechanical ventilation during admission. | 24 months
  Use of continuous positive airway pressure (CPAP) or biphasic positive airway pressure (BiPAP), mechanical ventilation during admission, as documented in patient's admission record.
Cardiac arrest | 24 months
  Whether the child experienced a cardiac arrest during their admission.
Death | 24 months
  Whether the child died during their admission.
Return visits | 24 months
  Using administrative data and parent surveys, we will measure return visits to the Emergency Department, and hospitalizations within 30 days following the initial bronchiolitis admission, overall and for respiratory illness.
Use of low-flow supplemental oxygen | 24 months
  Any use of low-flow supplemental oxygen, and duration of use.
Fluid supplementation | 24 months
  Presence and type (intravenous vs. nasogastric) of fluid supplementation
Nil per os order | 24 months
  Any order for "nil per os" (feeding not permitted) during admission.
Chest X-ray results | 24 months
  Results of chest X-rays ordered. Obtained from medical record.
Presence of bacterial co-infection | 24 months
  Presence and type of bacterial co-infections. Obtained from medical record.
Use of inhaled corticosteroids | 24 months
  Whether inhaled corticosteroids were administered during admission. Obtained from medical record.
Use of chest physiotherapy | 24 months
  Whether chest physiotherapy was performed during admission. Obtained from medical record.
Complete blood count | 24 months
  Results of complete blood count. Obtained from medical record. Numerical
Electrolyte levels | 24 months
  Electrolyte levels in blood. Obtained from medical record. Numerical
Venous blood gas | 24 months
  Results of blood tests ordered; venous blood gas. Obtained from medical record. Numerical
Antiviral prescription | 24 months
  Any prescription for an antiviral effective against influenza during admission.Obtained from medical record.
Prescription at discharge from hospital | 24 months
  Data collection on prescription at discharge from the hospital including the following: 1) repeat chest x-ray; 2) prescription for short-acting beta-agonists (SABA); 3) inhaled corticosteroids; 4) systemic corticosteroids; 5) antibiotics; and 6) antivirals.
Care received in the 30 days following discharge. | 24 months
  Care received in the 30 days following the patient's discharge from the hospital, including outpatient follow-up appointments in the following 30 days, follow-up chest x-rays, as well as prescription for antibiotics, short-acting beta-agonists, and inhaled corticosteroids.
Length of stay | 24 months
  Length of hospital stay in hours, both in the ED and inpatient unit, measured using recorded time of arrival and departure to and from the ED and inpatient unit.
Cost of hospitalization | 24 months
  Cost of hospitalization will be evaluated from a healthcare institution perspective with data from hospital decision support. More detailed costs data (micro-costing) will also be obtained whenever possible, allowing differentiation between services not readily discerned by traditional case costing methods typically based on resource intensity weights.
Use of Heated humidified high-flow nasal cannula (HHHFNC) | 24 months
  Heated humidified high-flow nasal cannula (HHHFNC) help reduce work of breathing and can be beneficial in severe bronchiolitis cases. We will measure proportion of HHHFNC use in hospitalized children with bronchiolitis stratified by disease severity. Obtained from medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Drouin, MD, MSc, MPH, Principal Investigator — CHU Sainte-Justine Research Centre
Locations (15):
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - Children's Hospital of Western Ontario (London Health Science Centre), London, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre hospitalier Cité-de-la-Santé, Laval, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier Université Laval - Centre Mère-Enfant Soleil, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No